CLINICAL TRIAL: NCT01554683
Title: Seizure-like Hippocampal Activity in Alzheimer's Disease Neurodegeneration
Brief Title: Seizure Activity in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Press, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011P000303
Record Dates: First submitted 2012-02-21; First posted 2012-03-15 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease; Seizures
Keywords: Alzheimer's Disease; Seizures; Memory; Executive
MeSH Terms: conditions — Alzheimer Disease; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Dose Levetiracetam (Active Comparator): Low Dose Levetiracetam administration via IV infusion over 20 min
  Interventions: Drug: Low/High/Placebo Dose Keppra (Levetiracetam)
- Low Dose Levetiracetam (Active Comparator): High Dose Levetiracetam administration via IV infusion over 20 min
  Interventions: Drug: Low/High/Placebo Dose Keppra (Levetiracetam)
- Placebo administration (Placebo Comparator): Saline administration via IV infusion over 20 min
  Interventions: Drug: Low/High/Placebo Dose Keppra (Levetiracetam)

INTERVENTIONS:
Drug: Low/High/Placebo Dose Keppra (Levetiracetam) — Low Dose (2.5 mg/kg) High Dose (7.5 mg/kg) Placebo (Saline)
  Other Names: Levetiracetam

SUMMARY:
The main purpose of this research project is to study how seizure-like activity affects the blood flow in the brain of patients with Alzheimer's disease (AD). Changes in blood flow can change memory and thinking ability, as happens in Alzheimer's disease. The investigators are using a study drug called Levetiracetam, which helps control seizure-like activity to see if it can help change the abnormal blood flow in the brain that is seen in some people with Alzheimer's disease.

DETAILED DESCRIPTION:
Subjects will make four separate visits to BIDMC. Subject will come to the Clinical Research Center. All of the visits will take around 5 hours apiece.

If subjects agree to be in this study, subjects will be asked to read and sign the consent form. After subjects sign the consent form, the following things will happen:

1. Screening Procedures: Screening procedures are tests and procedures that will be done to determine if subjects are eligible to take part in the research study. For this research study, the screening procedures include:

   * A thorough medical history. Investigators will ask if subjects have any medical problems. Investigators will ask about subjects Alzheimer's disease and if they have had any seizures.
   * A physical examination. Investigators will take your blood pressure and your heart rate. They will examine your heart and lungs and take your height and weight
   * Investigators will also assess the subject's nervous system. Investigators will examine subject's speech, memory, strength, coordination, and reflexes.
   * Investigators will ask you to take some paper and pencil tests. This will help us to understand your memory and mood
   * Subjects will have a blood test to check how your kidneys are functioning.

   Subjects may have already had some of these tests done by their doctor when they were diagnosed with Alzheimer's disease.

   The information we learned will help to decide whether subjects could join the study. Investigators will explain the reason if they decide subjects should not join the study. Our decision does NOT mean that subjects have a health problem or disorder .
2. Randomization Procedures: Investigators will meet with one of the study doctors if subjects continue in the study. The study doctor will explain to subjects when they are expected to come to the research center for study testing or to take the study drug. Subjects will come to the BIDMC Clinical Research Center for three visits. These visits will occur within one month.

   All study participants will receive the same study drugs over the three (3) visits.
   * Subjects will receive levetiracetam, the study drug, in a low dose, 2.5 milligrams for each kilogram of body weight, at one visit.
   * Subjects will receive levetiracetam, the study drug, in a high dose, 7.5 milligrams for each kilogram of body weight, at one visit.
   * Subjects will receive a placebo at one visit.

   A placebo is an inactive injection that looks like the study drug, but a placebo contains no active medication. In this study, the placebo is a saline (sterile salt water) injection.

   Sometimes study results are truly due to the study medication. Sometimes the study results are not due to the study medication. Investigators are using a placebo to help us understand the reason for the results in this study.

   The order of the above visits will not be the same for all study participants. There are six different orders to receive the study drugs. For example, subjects could receive the placebo at the first visit, the high dose of levetiracetam at the second visit, and the low dose of levetiracetam at the third visit. Another example is that subjects could receive the low dose at the first visit, the placebo at the second visit, and the high dose at the third visit.

   Deciding the order in which you get the study drugs will be done by to a method called "randomization." Randomization means that a computer will assign patients to study drugs in a random manner, like flipping a coin. Another way to say randomization is "by chance." When you flip a coin, you get heads or tails by chance. The chance of getting any dose of study drug or placebo is about equal. After the randomization, Subjects will be assigned to get one study drug or placebo at each visit. Subjects will not be able to choose which study drug you will get at each visit.

   Subjects will not know which study drug dose or placebo will be given at a visit. The study doctor will not know which study drug dose or placebo will be given at a visit. The study doctor can find out this information quickly if there is an emergency.
3. Research Procedures: Subjects will come to the BIDMC Clinical Research Center three times if they continue in this study. A member of the study team will meet subjects when they arrive. Subjects will first have an intravenous catheter (also called an IV) put into a vein. A nurse will check blood pressure and heart rate. Subjects will have a brief physical exam and a nervous system exam by a doctor

   Subjects will then have an electroencephalogram (EEG). An EEG gives investigators information about the nervous system - specifically the brain. Subjects will have their scalp cleaned with alcohol and small discs - called electrodes - placed on the scalp using gel. Then the head will be will be wrapped with gauze to. keep the discs from moving. The discs will be attached by wires to an EEG machine. The EEG machine will be at the bedside and will give investigators information about the electrical activity in the brain. Subjects will need to lie quietly with eyes closed during the one hour that the EEG machine is attached. Investigators will clean the gel from hair and skin when the EEG is over.

   Investigators will give subjects either levetiracetam -- the study drug -- or placebo while subjects are having EEG. Investigators will give subjects the study drug or placebo through the intravenous catheter ("IV") in the arm. This will take around 20 to 30 minutes. The subjects nurse will take the subject's blood pressure and heart rate two times while the study drug is being given to the subject and again after it is finished. The subject will note any side effects they have during this time and after.

   Subjects will then review what will happen during the MRI scan with the Investigator. The MRI study will be conducted at the Magnetic Resonance Imaging Center of the Department of Radiology at the Beth Israel Deaconess Medical Center.

   The MRI is a method of taking pictures of the brain and of the blood flow in the brain, using a large magnet and radio signals. Subjects will be asked to lie down on a platform that can be slid into the magnet. An MRI imaging coil, which is made from special wires that are covered in plastic, will be placed around the head. Foam pads will be placed around the head to limit head movement during the scan. During the scan, subjects will be asked to lie still on their back for about 45 to 60 minutes. They will hear a loud knocking or hammering noise while the MRI is taking pictures, but the process itself will be painless. They will be given disposable earplugs to use to help lessen the noise. During the procedure, subjects will be in constant contact with the MRI technician through an intercom. If at any time during the scan you feel too uncomfortable to continue, no matter what the reason, the study will be immediately stopped and subjects will be removed from the magnet (MRI Scanner).

   Subjects will return to the Clinical Research Center after the MRI. They will take a few pencil-and-paper tests for about one hour. These tests will tell the investigator about memory and mood. They will also learn about your attention skills. Investigators will also learn about the subjects= language skills and "handedness" (a tendency to favor right or left hand).

   As the medication (levetiracetam) may make the subject drowsy, they will not be able to drive. Someone will need to accompany them to and from the hospital for the three study visits.

   The second and third study visits will have the same sequence of events.

   SUMMARIES

   Here is a summary of the Screening Visit

   Screening visit / informed consent Review your medical history. Brief physical and neurological exam. Paper and pencil tests. Blood drawn to check the functioning of kidneys. Review and sign the informed consent form.

   Here are summaries of the three Study Visits

   Visit One

   :

   Vital signs. 2 minutes Brief physical and neurological exam. 10 minutes An intravenous catheter placed in your arm. 5 minutes EEG. 60 minutes Intravenous dose of the medication, levetiracetam, or placebo. 20 minutes MRI scan. 60 minutes Paper and pencil tests. 60 minutes

   Study Visit Two: (This visit will occur one to two (1-2 )weeks after Study Visit One)

   Vital signs. 2 minutes Brief physical and neurological exam. 10 minutes Intravenous catheter placed in your arm. 5 minutes EEG. 60 minutes Intravenous dose of the medication, levetiracetam, or placebo. 20 minutes MRI scan. 60 minutes Paper and pencil tests. 60 minutes

   Study Visit Three: (This visit will occur one to two (1-2 )weeks after Study Visit Two)

   Vital signs. 2 minutes Physical and neurological exam. 10 minutes Intravenous catheter placed in your arm. 5 minutes EEG. 60 minutes Intravenous dose of the medication, levetiracetam, or placebo. 20 minutes MRI scan. 60 minutes Paper and pencil tests. 60 minutes

   Each visit will take a total of approximately 5 hours. This includes the time for the EEG, MRI imaging and neuropsychological tests. Subjects will be allowed time to rest between activities on a bed if they become tired. The CRC staff will serve lunch.
4. Monitoring/Follow-Up Procedures. Procedures performed to evaluate the effectiveness and safety of the research procedures are called "monitoring" or "follow-up" procedures. Subject follow-up procedure will be a phone call from the study doctor one week after the third visit. They will ask if any side effects from the study or study medication occurred

Timing: If subjects are enrolled into the study following the initial screening visit, each of the three study visits will be separated by 2-3 week intervals. Therefore, the entire study will last approximately 6-9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meets the NINCDS-ADRDA criteria for probable Alzheimer's disease
* Mild AD (MMSE ≥ 20)
* Age >= 50 years
* English as first language

Exclusion Criteria:

* A history of seizures prior to the onset of AD
* Familial Alzheimer's Disease due to known genetic mutations
* Current use of an antiepileptic medication
* Current use of a medication known to lower seizure threshold (e.g. bupropion or a neuroleptic)
* Presence of parkinsonism
* Significant cerebrovascular disease
* Other Central Nervous System disease (e.g. stroke, severe traumatic brain injury)
* Major depression or other psychiatric or behavioral disorders (psychosis, agitation)
* Medical contraindication to MRI (e.g. pacemaker, intraocular or intracranial metallic objects)
* Severe claustrophobia or inability to lie flat for MRI
* Known allergy to levetiracetam, or history of previous adverse reaction to levetiracetam
* Serum creatinine >= 2
* A score of >9 on the Geriatric Depression Scale

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Press, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Berenson Allen Center Lab Website — http://tmslab.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: While 12 participants were consented, 3 withdrew prior to receiving medications. 2 were due to claustrophobia preventing MRI and one was due to inability to recall why they were doing the study (so study was discontinued prior to drug administration).
Groups:
- High Dose Levetiracetam, Low Dose, Placebo: levetiracetam given at a dose of 7.5mg/kg over 20 minutes followed by LEV at a dose of 2.5mg/kg over 20 minutes followed by Placebo over 20 minutes
- Low Dose Levetiracetam, High Dose, Placebo: Levetiracetam given at a dose of 2.5mg/kg over 20 minutes followed by LEV at 7.5mg/kg over 20 minutes followed by Placebo
- Placebo Administration, High Dose LEV, Low Dose: Saline administration via IV infusion over 20 min followed by LEV at 7.5mg/kg followed by LEV at 2.5 mg/kg
- High Dose LEV, Placebo, Low Dose: LEV at 7.5mg/kg followed by Placebo, followed by LEV at 2.5mg/kg
- Low Dose LEV, Placebo, High Dose LEV: Low dose LEV at 2.5mg/kg followed by placebo followed by High Dose LEV at 7.5mg/kg
- Placebo, Low Dose LEV, High Dose LEV: Placebo, followed by low dose LEV at 2.5mg/kg followed by High dose LEV at 7.5mg/kg
Period: Overall Study
Arm/Group | High Dose Levetiracetam, Low Dose, Placebo | Low Dose Levetiracetam, High Dose, Placebo | Placebo Administration, High Dose LEV, Low Dose | High Dose LEV, Placebo, Low Dose | Low Dose LEV, Placebo, High Dose LEV | Placebo, Low Dose LEV, High Dose LEV
Started | 2 | 1 | 3 | 2 | 1 | 0
Completed | 2 | 1 | 3 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Saline administration via IV infusion over 20 min, High dose LEV 7.5mg/kg, and Low dose LEV at 2.5mg/kg in random order
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Evaluable fMRI Scans
Description: Number of participants who had evaluable fMRI scans with arterial spin labeling to measure brain perfusion blood flow changes in specific brain regions, including the hippocampus
Time Frame: 3 MRIs acquired at visit 2,3 and 4 between weeks 1 and 6
Measure: Number; unit: participants
Groups:
- High Dose Levetiracetam: levetiracetam given at a dose of 7.5mg/kg over 20 minutes
- Low Dose Levetiracetam: Levetiracetam given at a dose of 2.5mg/kg over 20 minutes
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
Number analyzed (Participants) | 9 | 9 | 9
participants
  temporal lobe perfusion | 9 | 9 | 9
  Frontal lobe perfusion | 9 | 9 | 9

2. Secondary Outcome: Free and Cued Selective Reminding Test
Description: Evaluate memory changes, the free and cued selective reminding test lists the number of items recalled from a possibility of 16, adding free recall at two time points, yielding a score on a 0-32 scale per participant. A higher score is better, representing better recall.
Time Frame: At visits 2,3,4 in weeks 1-6 (one visit per intervention, visits spaced 2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
Number analyzed (Participants) | 9 | 9 | 9
score on a scale | 13.4 (10) | 14.3 (5.4) | 15 (8)

3. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: Evaluate AD severity, this is a 30 point scale from 0-30, with higher scores representing better performance.
Time Frame: At visits 2,3,4 in weeks 1-6 (*one visit per intervention, visits spaced 2 weeks apart
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
Number analyzed (Participants) | 9 | 9 | 9
score on a scale | 21.4 (1.7) | 21.4 (3) | 20.4 (4.1)

4. Secondary Outcome: Trial Making Test Parts A & B
Description: Evaluate visuo-spatial changes, outcome is total time to complete a task of connecting items (either numbers in trails A, or numbers alternating with letters in Trails B). A longer time indicates worse performance.
Time Frame: At visits 2,3,4 in weeks 1-6 (*one visit per intervention, visits spaced 2 weeks apart*
Measure: Geometric Mean (Standard Deviation); unit: seconds
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
Number analyzed (Participants) | 9 | 9 | 9
seconds
  Trails A | 44.1 (14.7) | 47.1 (25.9) | 48.9 (24.1)
  Trails B | 147.3 (44.4) | 138.9 (45.3) | 153.5 (64.1)

5. Secondary Outcome: Phonemic & Category Fluency Test
Description: Evaluate memory changes in AD. Phonemic fluency refers to the number of items generated in one minute beginning with a specific letter. A higher score indicates more items and better performance. There is no maximum score. Category fluency refers to the number of items generated belonging to a specific category (such as animals), again, more items generated indicates better performance.
Time Frame: At visits 2,3,4 in weeks 1-6 (*one visit per intervention, visits spaced 2 weeks apart*
Measure: Mean (Standard Deviation); unit: Correct Items
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
Number analyzed (Participants) | 9 | 9 | 9
Correct Items
  Phonemic fluency | 34.4 (12.5) | 34 (9.5) | 34.4 (13.2)
  Animal fluency | 13.4 (5.5) | 13.1 (3.7) | 12.4 (5.7)

ADVERSE EVENTS:
Time Frame: 6 weeks, from beginning of study to end of study (study consisted of 3 separate infusions, all side effects were assessed over the 6 hours after the infusions)
Arm/Group | High Dose Levetiracetam | Low Dose Levetiracetam | Placebo Administration
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT01554683/Prot_SAP_000.pdf